CLINICAL TRIAL: NCT02876874
Title: the Relationship Between the Activity of Rheumatoid Arthritis（RA） and Popliteal/Epitrochlear Lymph Node Morphology and the Drainage of Hand/Foot Superficial Lymphatic Vessels
Brief Title: Relationship Between the Activity of Rheumatoid Arthritis and Lymph Node Morphology and Lymphatics Drainage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RA and lymphatic vessels
Record Dates: First submitted 2015-02-03; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis; Lymph Node Mass; Lymphatic Vessel; Dilatation
Keywords: Rheumatoid Arthritis; lymph nodes morphology; drainage of lymphatic vessels
MeSH Terms: conditions — Arthritis, Rheumatoid; Dilatation, Pathologic | interventions — Indocyanine Green

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Peripheral blood 10ml for the analysis of cytokines,such as IL-1/6, TNF-α,VEGF-3 recepter,VEGFRC/E, et al.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- the patients group: 0.1ml, 5mg/ml indocyanine green(ICG) will be injected subcutaneously to aid visualization in NIR
  Interventions: Drug: indocyanine green(ICG)
- the health group: 0.1ml, 5mg/ml indocyanine green(ICG) will be injected subcutaneously to aid visualization in NIR
  Interventions: Drug: indocyanine green(ICG)

INTERVENTIONS:
Drug: indocyanine green(ICG) — ICG will be injected into the dorsal of hand/foot
  Other Names: IC-GREEN®(indocyanine green for injection,USP),AKORN,Inc

SUMMARY:
To observe the relationship between the activity of rheumatoid arthritis and popliteal/epitrochlear lymph node morphology and the drainage of hand/foot superficial lymphatic vessels

DETAILED DESCRIPTION:
Rheumatoid Arthritis patients and health participants will be recruited in our research. Then the classification of American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2009 will be used to identify rheumatoid arthritis patients. The measurement of disease activity are Disease Activity Score 28 (DAS28) combined with the synovitis, bone edema and bone erosion of hand and wrist detected by magnetic resonance (MR) and Doppler ultrasound (DUS).The morphology of lymph node in popliteal/epitrochlear are scanned by 3-dimensional MR and DUS. The drainage of hand/foot superficial lymphatic vessels are detected in sight of near infrared ray (NIR) with the applying of Indocyanine Green (ICG) subcutaneously. We'll conduct correlation analysis to reveal the relationship between the activity of Rheumatoid Arthritis and lymph nodes morphology and lymphatic vessels drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfilling the classification criteria of American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2009 (scores more than 6 points)
2. Health participants normal in the test of blood/urine/stool routine, liver and kidney functions, electrocardiogram and without obvious medical history
3. Age 18 to 65 years
4. Fulling understood the whole trial and written informed consent.

Exclusion Criteria:

Participants will be excluded when they combined with:

1. other types of autoimmune diseases such as ankylosing spondylitis, systemic lupus erythematosus, scleroderma, etc.,
2. lymphatic system disorders, such as lymphoma, lymphangitis and lymphatic edema due to lymphatic flow disorders,
3. disorders that effect the circulation of lymph or blood vessels such as hemangiomas,
4. tumors or cancer,
5. operation history within a year, such as joint orthopedics, tumor resection, etc.,
6. allergies or allergic to iodine, or radioactive iodine treatment within the last year,
7. with metal objects inside, such as pacemakers or nails,
8. the skin for the ultrasound inspection not intact such as eczema,ulceration, etc.,
9. lactation or pregnancy women or preparation to be pregnant within the next half year,
10. without whole limbs to inspect,
11. mania, depression or other mental disorder
12. medical disorders such as diabetes, hypertension or hyperlipidemia, etc.,
13. a history of infectious diseases such as tuberculosis, hepatitis B or HIV, etc.,
14. a history of drug abuse such as opioid analgesics, sedative-hypnotics or alcohol abuse, etc.,
15. severe liver or kidney dysfunction (Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) two times higher than the upper limit of normal, serum creatinine levels more than two times the upper limit of normal);
16. poor compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study conducted in Shanghai, China. The participants will be recruited by advertisement in in Longhua hospital, communities and universities in Shanghai.
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
T-initial | after the injection of ICG from the first day to the fourth day after
  the time that it takes for the ICG to be detected in vessels

SECONDARY OUTCOMES:
S-max | after the injection of ICG, 1day after, 2 days after, 3 days after and 4days after
  the maximum ICG signal intensity observed in the target lymph node during the first day imaging session
T-max | after the injection of ICG, 1day after, 2 days after, 3 days after and 4days after
  the time it takes for a nodes in cubital fossa or popliteal space to achieve maximal ICG signal intensity
%Clearance | after the injection of ICG, 1day after, 2 days after, 3 days after and 4days after
  an assessment of ICG wash out through the lymphatics and is quantified as the percent difference of ICG signal intensity between the two ICG-NIR images from a certain region at a) S-max (first day) and b) 24 hours post ICG injection,
Pulse | after the injection of ICG, 1day after, 2 days after, 3 days after and 4days after
  ICG pulses that pass the a certain region within 400 seconds.
lymphatic node size | the second day after enrollment
lymphatic node shape | the second day after enrollment
lymphatic node transverse/longitudinal diameter ratio | the second day after enrollment
lymphatic node types of edges | the second day after enrollment
lymphatic node thickness of cortex/medulla | the second day after enrollment
lymphatic node homogeneity | the second day after enrollment
lymphatic node hilum | the second day after enrollment
lymphatic node blood flow signal | the second day after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Yong-jun Wang, Dr., Principal Investigator — Longhua Hospital
Locations (2):
- China (2):
  - Longhua Hospital, Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Longhua Hospital, Shanghai University of TCM, Shanghai

IPD SHARING:
Plan to Share IPD: No